CLINICAL TRIAL: NCT06057285
Title: Efficacy of an Augmented Reality Application Developed for ACLs Training on the Knowledge and Skill Levels of Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A-ER-109-383
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: ACLs Learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR technologies to develop a first aid cart learning system (No Intervention): The control group received traditional teaching.
- An ACLs cart training course was developed using augmented reality (AR) technologies (Experimental): The developed first aid cart learning system was applied to ACLs drills in a regular ACLs training program, and an AR group used this learning system to assist in their learning. The AR group scanned the dedicated AR marker using a mobile device
  Interventions: Device: An ACLs cart training course was developed using augmented reality (AR) technologies

INTERVENTIONS:
Device: An ACLs cart training course was developed using augmented reality (AR) technologies — The developed first aid cart learning system was applied to ACLs drills in a regular ACLs training program, and an AR group used this learning system to assist in their learning. The AR group scanned the dedicated AR marker using a mobile device
  Arms: An ACLs cart training course was developed using augmented reality (AR) technologies

SUMMARY:
Background: Having Advanced Cardiac Life Support (ACLs) skills is essential for nurses. During the COVID-19 pandemic, augmented reality (AR) technologies were incorporated into medical education to increase learning motivation and accessibility.

Objectives: To determine whether using augmented reality for educational applications can significantly improve first aid cart learning, learning motivation, cognitive load, and system usability among nurses in ACLs training of nurses.

Design: The present study was a quasi-experiment study. Settings: The research setting was a medical center in southern Taiwan Participants: In total, 102 nurses completed the course, with 43 nurses in the AR group and 59 nurses in the control group.

Methods: An ACLs cart training course was developed using augmented reality (AR) technologies in the first stage. However, the efficacy of the developed ACLs training course was evaluated.

DETAILED DESCRIPTION:
Application Augmented Reality for ACLs training of Registered Nurse

ELIGIBILITY:
Inclusion Criteria: Nurses who were aged 20 years or older, could speak and read Mandarin, and completed the questionnaire after the research objective was explained were recruited.

Exclusion Criteria: Nurses without mobile devices were excluded.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
ACLs learning outcomes | one hour
  knowledge improve

CONTACTS AND LOCATIONS:
Locations (1):
- Wan-Na Sun, Tainan, no-US, Taiwan

REFERENCES:
- [Derived] Sun WN, Hsieh MC, Wang WF. Nurses' Knowledge and Skills After Use of an Augmented Reality App for Advanced Cardiac Life Support Training: Randomized Controlled Trial. J Med Internet Res. 2024 Dec 5;26:e57327. doi: 10.2196/57327. PMID 39636667